CLINICAL TRIAL: NCT04526808
Title: Effects of Low FODMAP Diet on Leaky Gut and Mucosal Immune Cell Abundance in Diarrhea-predominant Irritable Bowel Syndrome
Brief Title: Effects of Low FODMAP Diet on Leaky Gut
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, Judy Nee, Assistant Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2019P000149
Record Dates: First submitted 2020-08-05; First posted 2020-08-26 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — FODMAP Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FODMAP diet (Experimental)
  Interventions: Other: FODMAP diet

INTERVENTIONS:
Other: FODMAP diet — low FODMAP diet

SUMMARY:
The pathophysiology of Irritable bowel syndrome (IBS) is multifactorial involving complex interplay of altered intestinal permeability, mucosal immune activation, visceral hypersensitivity and gut dysbiosis. Although the exact triggers for these pathological changes in IBS are not clear but diet might play an important role. In fact, several studies have reported improvement in gastrointestinal symptoms on a diet low in FODMAPs (LFD) in patients with IBS, specifically in diarrhea predominant IBS (IBS-D). However, the mechanism of action of LFD is not well understood.

DETAILED DESCRIPTION:
we aim to evaluate the following in patients with IBS-D. The effect of LFD on colonic permeability. 2.The effect of LFD on abundance of colonic mucosal immune cells specifically T-cell and mast cell abundance 3.The effect of LFD on colonic mucosal microbiome

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65 years at the time of screening
* normal serum studies including serum tissue-transglutaminase antibodies, thyroid stimulating hormone levels, C-reactive protein, complete blood count since the onset of symptoms
* normal stool studies including C diff testing, culture, ova and parasites since the onset of symptoms
* IBS-SSS score of ≥175 at the end of 7-day screening period

Exclusion criteria:

* individuals already on a LFD or other dietary restriction such as gluten free diet within the past 6 months
* individuals with any known food allergy or insulin-dependent diabetes
* known history of celiac disease, inflammatory bowel disease or microscopic colitis
* prior small bowel or colonic surgery or cholecystectomy
* pregnant patients
* antibiotics in the past 3 months
* those who regularly use mast cell stabilizers or anti-histaminic or non-steroidal anti-inflammatory agents (NSAIDs) excluding daily baby aspirin or steroids or bile-acid binder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
colonic permeability | 4 weeks
  Lactulose:Mannitol ratio pre and post treatment

SECONDARY OUTCOMES:
colonic immune cells | 4 weeks
  expression of tight junction proteins pre and post treatment using RT-PCR
colonic microbiome | 4 weeks
  relative stool microbial abundance pre and post treatment measured using 16s RNA

CONTACTS AND LOCATIONS:
Overall Officials: Judy Nee, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No